CLINICAL TRIAL: NCT02419625
Title: The Epidemiology of Hepatitis E Virus Infection in Israel and Potential Risk Factors, a Multicenter, Comparative, Cross-sectional Study
Brief Title: The Epidemiology of Hepatitis E Virus Infection in Israel and Potential Risk Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eli Zuckerman, head of liver unit, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CMC-15-0021-CTIL
Record Dates: First submitted 2015-03-22; First posted 2015-04-17 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Hepatitis E
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- subgroup-specific HEV in Israel (Other): The study will involve patient interviews using questionnaires
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — questionnaires , serum samples will be used

SUMMARY:
Hepatitis E virus is a single-stranded positive-sense RNA virus with genome of approximately 7.2kb in length. The HEV genome is capped at the 5' end followed by a small untranslated region of 27 nucleotides and polyadenalated at the 3' end preceded by another UTR of 65 nucleotides . HEV has three open reading frames: ORF1, ORF2 and ORF3 that encode structural and non- structural proteins. ORF1 is the largest one, approximately 5,000 nt in length, located at the 5 ' end and encodes important proteins for the replication process (methyltransferase, papain-like cysteine protease, helicase, and RNA-dependent RNA polymerase). A noncoding, hypervariable region within ORF1 displays substantial genetic diversity; this region seems to modulate the efficiency of HEV replication. Notably, the differences in the genome size among different HEV strains are confined mainly to this region .ORF2 is located at the 3' end, encodes structural capsid proteins of 660 amino acids and contains three potential glycosylation sites. The ORF2 protein contains multiple immunogenic sites and neutralizing antibodies are directed against it al., .The essential region in the protein for immunogenicity is 452aa-617aa and the neutralizing epitopes have recently been shown to be conformational .ORF3 is located between the other two reading frames and encodes a small phosphoprotein of 123 amino acids. Its exact function has not been yet determined, however, multiple functions have been proposed. It is thought to interact with cellular mitogen-activated protein kinase phosphatase and other extracellular kinases, promoting cell survival through activation of intracellular signaling pathways .Moreover, the binding of the ORF3 encoded protein to host-specific proteins seems to influence the pathogenesis of HEV infections .A schematic drawing of the HEV genome is described in Figure 1 .

DETAILED DESCRIPTION:
General aim To identify the overall and subgroup-specific HEV sero-prevalence in Israel and examine associations between HEV seropositivity and putative risk factors.

3.2 Specific aims

* To determine the sero-prevalence of Israeli healthy population.
* To quantify the sero-prevalence of HEV infections in Israeli healthy population by age, gender, ethnicity, religion.
* To present the seroprevalence in five specific groups (farmers and swine veterinaries, unexplained acute hepatitis, immunosuppressed transplant recipients, immunosuppressed HIV patients) and identify if these specific population groups are at high risk of HEV sero-prevalence.
* To identify risk factors associated with an increased risk of HEV sero-prevalence in immunosuppressed transplant patients.
* To identify risk factors associated with an increased risk of HEV sero-prevalence in farmers and swine veterinaries.
* To identify the molecular characteristic of HEV in Israel and investigate the similarities to previously published HEV sequences.
* To identify the incidence of HEV seroconversion/ infection in transplant recipients. (sero-negative pre-transplanted patients will be tested consistently for HEV Ab's and HEV RNA after transplantation)

ELIGIBILITY:
* Patients who are followed-up in Carmel, Lin or Rambam Medical Centers who fulfill one or more of the following criteria and are willing to sign an inform consent
* Patients with elevated liver enzymes of unknown etiology
* Patients with acute hepatitis of unknown etiology
* Patients with chronic infection with hepatitis B , D or C.
* Immunosuppressed patients: patients with solid or haemato-oncologic malignancy or patients with chronic HIV infection.
* Patients with chronic liver disease of unknown etiology
* Participants who have contacts with swines: delivery, feeding, slaughtering, treatment)
* Healthy volunteers.

Inclusion criteria:

1. Patients with elevated liver enzymes of unknown etiology
2. Patients with acute hepatitis of unknown etiology
3. Patients with chronic infection with hepatitis B , D or C.
4. Immunosuppressed patients: patients with solid or haemato-oncologic malignancy or patients with chronic HIV infection.
5. Patients with chronic liver disease of unknown etiology
6. Participants who have contacts with swines: delivery, feeding, slaughtering, treatment)
7. Healthy volunteers.

Exclusion criteria:

1. Participants who do not fill the above criteria
2. Participants who are not willing to sign an inform consent
3. Participants younger than 18 year old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
study will measure the frequency of HEV infection in immune compromised population and in subjects with unexplained elevation of liver enzymes | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: eli zuckerman, Principal Investigator — Carmel Medical Center